CLINICAL TRIAL: NCT01699009
Title: A Nutritional Intervention for Migraines-2
Acronym: WCCR-MIG2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: WCCR-MIG2
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2014-05

CONDITIONS: Migraines
Keywords: Migraines, diet, vegan, vegetarian, plant-based
MeSH Terms: conditions — Migraine Disorders | interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vegan diet (Experimental): The diet group will be asked to follow a low-fat, vegan diet for 16 weeks.
  Interventions: Other: Plant based diet
- Supplement group (Placebo Comparator): The supplement group will follow an unrestricted diet, but will be given a pill containing a small, clinically insignificant amount of omega- 3 oils and vitamin E, which will serve as a placebo.
  Interventions: Other: an unrestricted diet

INTERVENTIONS:
Other: Plant based diet
  Arms: Vegan diet
Other: an unrestricted diet
  Arms: Supplement group

SUMMARY:
The purpose of the study is to assess whether, in individuals with migraines, a low-fat, vegan diet improves pain more effectively than a control supplement or a placebo. The principal measures are pain as measured by Visual Analog Scale (VAS) and the change in migraines frequency. The study duration is 36 weeks.This study also tests that a low fat, plant-based (vegan) diet free of foods commonly identified as triggers improves mood, using the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R), and the Beck Depression Inventory II (BDI-II).

DETAILED DESCRIPTION:
Preliminary evidence suggests that low-fat, vegetarian diets and certain nutritional supplements can help reduce pain and also reduce the need for pain medications for some people. The investigators will ask about 100 people to participate. All of them will get a low-fat, vegan diet and a nutritional supplement (mixture of omega-3 oils and vitamin E or a placebo), although some will get the diet first, and others will get the supplement first. This order in which they will get the diet and the supplement will be determined randomly, that is, by chance (like the toss of a coin). The principal measures are pain as measured by Visual Analog Scale (VAS)and the change in migraines frequency.

Mood change will be measured using the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R), and the Beck Depression Inventory II (BDI-II).

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of migraine, as defined by the criteria of the second edition of the International Classification of Headache Disorders:

At least 5 attacks fulfilling criteria the criteria below:

* Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)
* Headache has at least two of the following characteristics:
* unilateral location
* pulsating quality
* moderate or severe pain intensity
* aggravation by or causing avoidance of routine physical activity (eg, walking or climbing stairs)
* During headache at least one of the following:
* nausea and/or vomiting
* photophobia and phonophobia Not attributed to another disorder
* Migraines occurring at least twice per month, on average.
* Age at least 18 years
* Ability and willingness to participate in all components of the study
* Willingness to be assigned to either the diet group or supplement group
* Migraine medications unchanged within last 6 weeks.

Exclusion Criteria:

* < 18 years of age
* Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
* Use of recreational drugs in the past 6 months (past drug use, if fully recovered, is not a criteria for exclusion)
* Pregnancy
* Unstable medical or psychiatric illness
* Likely to be disruptive in group sessions (as determined by research staff)
* Already following a low-fat, vegan diet
* Lack of English fluency
* Inability to maintain current medication regimen
* Inability or unwillingness to participate in all components of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Migraines Pain Change in Migraines frequency | Baseline and 4 months
  Pain as measured by VAS score
Change in Migraines frequency | Baseline and 4 months
  the reduction in the number of migraine attacks.
Improvement in Mood | Baseline and 4 months
  mood changes will be measured using the Beck Depression Inventory II (BDI-II).
Improvement in Mood | Baseline and 4 months
  Mood changes will be measured using the Center for Epidemiologic Studies Depression Scale-Revised (CESD-R).

SECONDARY OUTCOMES:
Quality of life | Baseline and 4 months
  Health related quality of life as measured by a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, MD, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Bunner AE, Agarwal U, Gonzales JF, Valente F, Barnard ND. Nutrition intervention for migraine: a randomized crossover trial. J Headache Pain. 2014 Oct 23;15(1):69. doi: 10.1186/1129-2377-15-69. PMID 25339342